CLINICAL TRIAL: NCT07339644
Title: Functional Lung Avoidance Radiotherapy Guided by 4DCT Pulmonary Ventilation Function Imaging: A Prospective Single-arm Clinical Study
Acronym: 4DCT-FLAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, ZhenZhou Yang, Professor of Radiation Oncology, Cancer Center, Second Affiliated Hospital of Chongqing Medical University, The Second Affiliated Hospital of Chongqing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-2025-243
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer (Including Metastatic Cancer); Radiation Pneumonitis; Radiation-induced Lung Injury
Keywords: Functional lung avoidance radiotherapy; 4DCT ventilation imaging; Functional lung imaging (FLI); Dose-volume histogram (DVH); High-function lung; Radiotherapy planning optimization; Radiation pneumonitis; Pulmonary function
MeSH Terms: conditions — Lung Neoplasms; Radiation Pneumonitis

STUDY DESIGN:
Intervention Model Description: Single-arm, single-center prospective study. All participants receive 4DCT ventilation imaging-guided functional lung avoidance radiotherapy (FLAR). For within-patient paired dosimetric comparison, a conventional anatomic plan (non-functional plan) is also generated for each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 4DCT-FLI-Guided Functional Lung Avoidance Radiotherapy (FLAR) (Experimental): Participants receive IMRT planned with 4DCT ventilation functional imaging guidance. A ventilation map is generated from 4DCT, high-function lung (top 80% ventilation) is contoured, and the treatment plan is optimized to spare high-function lung while maintaining target coverage and meeting standard OAR constraints. A conventional anatomic plan is also generated for within-patient dosimetric comparison.
  Interventions: Procedure: 4DCT Ventilation Imaging-Guided Functional Lung Avoidance Radiotherapy (FLAR)

INTERVENTIONS:
Procedure: 4DCT Ventilation Imaging-Guided Functional Lung Avoidance Radiotherapy (FLAR) — All participants undergo 4DCT simulation. A ventilation map is generated from 4DCT data, and the high-function lung is defined as the top 80% ventilation region. This structure is imported into the treatment planning system, and an IMRT plan is optimized to preferentially spare high-function lung while maintaining target (PTV) coverage and meeting standard organ-at-risk constraints. A conventional anatomic plan (without functional guidance) is also created for within-patient paired dosimetric comparison.
  Other Names: Functional Lung Avoidance Radiotherapy; 4DCT-FLAR; 4DCT Ventilation Functional Imaging (4DCT-FLI)-Guided Radiotherapy

SUMMARY:
This prospective, single-center, single-arm study will evaluate the feasibility and safety of 4DCT ventilation functional imaging-guided functional lung avoidance radiotherapy (FLAR) in patients with lung malignancies receiving IMRT radiotherapy.

All participants will undergo 4DCT simulation as part of routine radiotherapy preparation. A ventilation map will be generated from 4DCT data, and the top 80% ventilation region will be defined as the high-function lung. This structure will be imported into the treatment planning system to create an FLAR plan that prioritizes sparing of high-function lung while maintaining target coverage (PTV D95%) and meeting standard dose constraints for organs at risk. A conventional anatomic plan (without functional guidance) will also be created for paired, within-patient dosimetric comparison.

The primary outcome is improvement in dosimetric sparing of the high-function lung (V10, V20, V30, and mean lung dose). Secondary outcomes include the incidence of grade ≥2 radiation pneumonitis (CTCAE v5.0), changes in pulmonary function (e.g., FEV1 and DLCO), and lung-related quality-of-life scores. Assessments will be performed mid-treatment (after 15 fractions), at the end of radiotherapy (after 30 fractions), and at 1, 3, 6, and 12 months after radiotherapy. The study plans to enroll 100 participants and follow each participant for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 85 years (inclusive); any sex.
* Diagnosed lung malignancy requiring thoracic radiotherapy (e.g., non-small cell lung cancer, small cell lung cancer, or pulmonary metastases).
* Planned to receive thoracic radiotherapy using either conventionally fractionated IMRT/VMAT or stereotactic body radiotherapy (SBRT), and able to complete pre-treatment 4DCT simulation suitable for generating a ventilation map.
* Adequate baseline organ function and clinically judged able to tolerate radiotherapy; ECOG performance status 0-1.
* No absolute contraindication to pulmonary function testing; patients with moderate COPD or impaired lung function may be included if the treating team judges radiotherapy to be tolerable.
* Able to comply with treatment and follow-up assessments.
* Written informed consent provided.

Exclusion Criteria:

* Pregnant or breastfeeding women. Women of childbearing potential must have pregnancy excluded prior to radiotherapy per institutional practice.
* Age <18 or >85 years.
* Uncontrolled severe cardiopulmonary disease or other severe comorbidities that make radiotherapy excessively high risk (e.g., decompensated heart failure, unstable cardiopulmonary status, active severe pulmonary infection).
* Prior high-dose thoracic radiotherapy to the same region such that safe re-irradiation is not feasible.
* Concurrent other active/advanced malignancy requiring priority treatment that would confound study outcomes.
* Recent participation in another interventional clinical trial or concurrent investigational therapy judged likely to interfere with this study's endpoints.
* Severe psychiatric, cognitive, or other conditions that prevent cooperation with radiotherapy and/or scheduled follow-up.
* Inadequate 4DCT image quality or inability to generate/validate the 4DCT ventilation map required for functional-lung-guided planning.
* Any other condition deemed unsuitable by the investigators in the interest of participant safety.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-24 (Actual); Primary Completion 2026-12-24 (Estimated); Study Completion 2027-12-24 (Estimated)

PRIMARY OUTCOMES:
Incidence of Radiation-Induced Lung Injury (Grade ≥2) | Time Frame: Assessed at 3 months, 6 months, and 12 months after completion of radiotherapy.
  Incidence of radiation-induced lung injury (RILI) of Grade ≥ 2, assessed using the Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0.
  CTCAE grades range from Grade 1 (mild) to Grade 5 (death related to adverse event), with higher grades indicating more severe toxicity.
  The primary outcome is the proportion of patients experiencing CTCAE Grade ≥ 2 RILI.

SECONDARY OUTCOMES:
Mean Dose to High-Function Lung (Gy) | At baseline treatment planning (prior to radiotherapy delivery).]
  DVH-derived mean dose to ventilation-defined high-function lung on paired plans (functional-lung-avoidance vs conventional plans). Lower dose indicates better sparing.
MLD for Whole Lung (Gy) | At baseline treatment planning (prior to radiotherapy delivery).
  Percentage volume (%) of ventilation-defined high-function lung receiving ≥5 Gy, reported separately for functional-lung-avoidance and conventional radiotherapy plans.
V5 of High-Function Lung (%) | At baseline treatment planning (prior to radiotherapy delivery).
  Percentage volume (%) of ventilation-defined high-function lung receiving ≥5 Gy, reported separately for functional-lung-avoidance and conventional radiotherapy plans.
V20 of High-Function Lung（%） | At baseline treatment planning (prior to radiotherapy delivery).
  DVH-derived V20 of ventilation-defined high-function lung, defined as the percentage of lung volume receiving ≥20 Gy, compared between functional-lung-avoidance and conventional radiotherapy plans.
Mean Dose to Heart (Gy) | At treatment planning (baseline, pre-radiotherapy delivery).
  DVH-derived mean dose (Dmean) to the heart, compared between functional-lung-avoidance and conventional radiotherapy plans.
Maximum Dose to Esophagus (Gy) | At treatment planning (baseline, pre-radiotherapy delivery).]
  DVH-derived maximum dose (Dmax) to the esophagus, compared between functional-lung-avoidance and conventional radiotherapy plans.
Maximum Dose to Spinal Cord (Gy) | At treatment planning (baseline, pre-radiotherapy delivery).
  DVH-derived maximum dose (Dmax) to the spinal cord, compared between functional-lung-avoidance and conventional radiotherapy plans.
Target Coverage (PTV D95) | At treatment planning (baseline, pre-radiotherapy delivery).
  Percentage of planning target volume (PTV) receiving at least 95% of prescribed dose, compared between functional-lung-avoidance and conventional plans.
Conformity Index of Radiotherapy Plans | At treatment planning (baseline, pre-radiotherapy delivery).
  Conformity Index (CI) of paired treatment plans, comparing functional-lung-avoidance and conventional anatomic radiotherapy plans.
  The Conformity Index is defined as the ratio of the prescription isodose volume to the target volume (CI = VRI / VT).
  The score ranges from 1.0 to >2.0, where a value closer to 1.0 indicates better conformity and thus higher plan quality.
Homogeneity Index of Radiotherapy Plans | At treatment planning (baseline, pre-radiotherapy delivery).
  Homogeneity Index (HI) of paired treatment plans, comparing functional-lung-avoidance and conventional anatomic radiotherapy plans.
  The Homogeneity Index is defined as (D2% - D98%) / D50%.
  The score typically ranges from 0 to 1.0, where lower values indicate more homogeneous dose distribution and better plan quality.
Gradient Measure (GM) of Radiotherapy Plans | At treatment planning (baseline, pre-radiotherapy delivery).
  Gradient Measure (cm) of paired radiotherapy plans, comparing 4DCT-FLI-guided functional lung avoidance plans and conventional anatomic plans. GM is defined as the difference between the equivalent sphere radii of the 50% and 100% prescription isodose volumes (GM = R50% - R100%); lower values indicate steeper dose fall-off and better plan quality.
Forced Expiratory Volume in 1 Second (FEV1) | Baseline and 1, 3, 6, and 12 months after radiotherapy.
  FEV1 measured by standardized spirometry (L and % predicted). Outcome is change from baseline.
Diffusing Capacity of the Lung for Carbon Monoxide (DLCO) | Baseline and 1, 3, 6, and 12 months after radiotherapy.
  DLCO measured using a standardized single-breath method (mL/min/mmHg and % predicted). Outcome is change from baseline.
Forced Vital Capacity (FVC) | Baseline and 1, 3, 6, and 12 months after radiotherapy.
  FVC measured by standardized spirometry (L and % predicted). Outcome is change from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: zhengjun Guo, MD., Principal Investigator — The Second Clinical College of Chongqing Medical University: The Second Affiliated Hospital of Chongqing Medical University
Locations (1):
- Cancer Center, Second Affiliated Hospital of Chongqing Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mattila S, Sovijarvi AR, Harjula A, Viljanen A, Takkunen O, Takkunen H, Mattila I, Mattila P, Merikallio E. Effects of mitral valve replacement on ventilation, volumes, diffusing capacity and regional perfusion of lungs in patients with mitral valve disease. Ann Chir Gynaecol. 1985;74(2):82-5. PMID 3875308